CLINICAL TRIAL: NCT04179500
Title: An Open-Label Phase 2 Trial to Evaluate the Male Reproductive Safety of a 6-Month Combination Treatment for Pulmonary Tuberculosis (TB) of Bedaquiline Plus Pretomanid Plus Moxifloxacin Plus Pyrazinamide (BPaMZ) in Adult Male Participants With Drug Resistant Pulmonary TB
Brief Title: A Trial to Evaluate the Male Reproductive Safety of Pretomanid in Adult Male Participants With Drug Resistant Pulmonary Tuberculosis
Acronym: PaSEM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pa-824-CL-012
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-09

CONDITIONS: Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant; Tuberculosis, MDR; Tuberculosis; Drug-Resistant Tuberculosis
Keywords: tuberculosis; TB; DR-TB; pretomanid (PA); PA-824; XDR TB; Pa
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant; Tuberculosis; Extensively Drug-Resistant Tuberculosis | interventions — pretomanid; bedaquiline; Moxifloxacin; Pyrazinamide

STUDY DESIGN:
Intervention Model Description: Phase 2 single arm multi-center, open-label clinical trial in DR-TB participants. Participants will receive bedaquiline 200 mg once daily for 8 weeks then 100 mg once daily for 18 weeks together with pretomanid 200 mg
  + moxifloxacin 400 mg + pyrazinamide 1500 mg once daily (BPaMZ) for 26 weeks.
  Participants will be followed for 52 weeks after end of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Participants (Experimental): Participants will receive bedaquiline 200 mg once daily for 8 weeks then 100 mg once daily for 18 weeks together with pretomanid 200 mg + moxifloxacin 400 mg + pyrazinamide 1500 mg once daily (BPaMZ) for 26 weeks.
  Interventions: Drug: Pretomanid; Drug: Bedaquiline; Drug: moxifloxacin; Drug: pyrazinamide

INTERVENTIONS:
Drug: Pretomanid — pretomanid 200 mg (once daily) for 26 weeks (with meal)
  Other Names: Pa-824; Doprevla; Pa
Drug: Bedaquiline — bedaquiline 200 mg (once daily) for 8 weeks (with meal), then bedaquiline 100mg (once daily) for 18 weeks (with meal)
  Other Names: Sirturo; B
Drug: moxifloxacin — moxifloxacin 400 mg (once daily) for 26 weeks (with meal)
  Other Names: Avelox; M
Drug: pyrazinamide — pyrazinamide 1500 mg (once daily) for 26 weeks (with meal)
  Other Names: Pyzina; Tebrazid; Z

SUMMARY:
Pretomanid is being used in an antimicrobial combination regimen(s) to treat patients with pulmonary tuberculosis (TB). The primary purpose of the Male Reproductive Safety - "BPaMZ/SEM"- clinical study is to evaluate the potential effect of pretomanid on human testicular function whilst being used in a 26 weeks antimicrobial combination regimen consisting of bedaquiline (B) plus pretomanid (Pa) plus moxifloxacin (M) and pyrazinamide (Z) (BPaMZ).

DETAILED DESCRIPTION:
The primary objective of this study is to assess the male reproductive safety of pretomanid in the regimen (BPaMZ) of bedaquiline 200mg (200mg daily for 8 weeks then 100 mg daily for 18 weeks), together with pretomanid 200 mg (1x daily) + moxifloxacin 400 mg (1x daily) + pyrazinamide 1500 mg (1 x daily) for 26 weeks in participants with drug-resistant pulmonary tuberculosis (DR-TB).

The secondary objective of the study is to evaluate the tuberculosis (TB) treatment efficacy, safety and tolerability after 26 weeks of active treatment for TB and follow up until 52 weeks after end of the above-described treatment regimen in participants with DR-TB.

ELIGIBILITY:
Inclusion Criteria:

1. Understands study procedures and voluntarily provides written informed consent prior to the start of any study-specific procedures.
2. Male gender 18 years or over
3. Body weight (in light clothing and no shoes) ≥ 45kg.
4. A positive molecular test for tuberculosis in sputum either at screening or within one month prior to enrolment.
5. Disease Characteristics:

   * Participants must have been diagnosed with TB prior to or at screening
   * Participants' TB should be resistant to rifampicin and/or isoniazid, and susceptible to fluoroquinolones by rapid sputum-based tests.
   * Participants who have had previous treatment for DR-TB for more than 3 months at start of screening should be discussed with the medical monitor.
6. A chest x-ray, within 26 weeks prior to or at the screening visit, which in the opinion of the Investigator is compatible with pulmonary TB

Exclusion criteria:

1. Resistant to fluoroquinolones by rapid molecular test
2. History of male infertility or vasectomy
3. Unable to produce semen sample
4. Evidence at screening of azoospermia
5. Known erectile dysfunction that would prevent ejaculation.
6. Historical or active disease process of the male reproductive tract that would compromise sperm production. e.g. tuberculous epididymitis.
7. History of any illness that, in the opinion of the Investigator, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
8. For HIV infected participants any of the following:

   1. CD4+ count <100 cells/μL
   2. Received intravenous antifungal medication within the last 90 days
9. Participants with newly diagnosed tuberculosis and HIV that require initiation of appropriate HIV therapy before participants has received at least 2 weeks of an antituberculosis regimen.
10. Received pretomanid and/or delamanid to treat TB
11. Known chronic hepatitis B or C
12. For HIV infected participants:

    1. The following antiretroviral therapy (ART) should not be used:

1. Stavudine 2. Zidovudine 3. Didanosine 4. Triple NRTI regimen is not considered optimal for HIV treatment (poor efficacy)

13. Participants with the following toxicities at screening as defined by the enhanced Division of Microbiology and Infectious Disease (DMID) adult toxicity table (Draft November 2007) where applicable:

1. Platelets <75,000/mm3
2. Creatinine >1.5 times upper limit of normal (ULN)
3. eGFR ≤ 60 mL/min
4. Haemoglobin <8.0 g/dL
5. Serum potassium less than the lower limit of normal for the laboratory. This may be repeated once
6. AST:

   * ≥3.0 x ULN to be excluded
   * results between 1.5 x ULN and 3 x ULN must be discussed with and approved by the Sponsor Medical Monitor
7. ALT:

   * ≥3.0 x ULN to be excluded
   * greater than ULN must be discussed with and approved by the Sponsor Medical Monitor
8. ALP:

   * ≥3.0 x ULN to be excluded
   * 2.0 - <3.0 x ULN must be discussed with and approved by the Sponsor Medical Monitor
9. Total bilirubin:

   * >1.5 x ULN to be excluded
   * Greater than ULN must be discussed with and approved by the Sponsor Medical Monitor
10. Direct bilirubin:

    • greater than 1x ULN to be excluded
11. Positive hepatitis B surface Ag, or hepatitis C antibody

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — males 18 years of age or older
Enrollment: 26 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2024-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lombardi, MD, Study Chair — Global Alliance for TB Drug Development
Locations (4):
- National Center for Tuberculosis and Lung Diseases, Tbilisi, Georgia
- South Africa (3):
  - CHRU, Sizwe Tropical Diseases Hospital, Johannesburg
  - Isango Lethemba TB Research Unit Empilweni TB Hospital, Port Elizabeth
  - The Aurum Institute: Rustenburg Clinical Research Centre, Rustenburg

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No pre-assignment events occurred.
Groups:
- BPaMZ: Participants will receive bedaquiline 200 mg once daily for 8 weeks then 100 mg once daily for 18 weeks together with pretomanid 200 mg + moxifloxacin 400 mg + pyrazinamide 1500 mg once daily (BPaMZ) for 26 weeks.
  Pretomanid: pretomanid 200 mg (once daily) for 26 weeks (with meal)
  Bedaquiline: bedaquiline 200 mg (once daily) for 8 weeks (with meal), then bedaquiline 100mg (once daily) for 18 weeks (with meal)
  moxifloxacin: moxifloxacin 400 mg (once daily) for 26 weeks (with meal)
  pyrazinamide: pyrazinamide 1500 mg (once daily) for 26 weeks (with meal)
Period: Treatment
Arm/Group | BPaMZ
Started | 26
Completed | 22
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 2
Not completed — pyrazinamide resistance | 1
Period: Follow-up
Arm/Group | BPaMZ
Started | 22
Completed | 18
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Total Enrolled
Arm/Group | BPaMZ
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  South Africa | 18
  Georgia | 8
Height [Mean (Standard Deviation); unit: cm] | 175.8 (7.3)
Weight [Least Squares Mean (Standard Deviation); unit: kg] | 62.2 (11.7)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 20 (3)
HIV Status [Count of Participants; unit: Participants]
  Positive | 8
  Negative | 18
Smoking [Count of Participants; unit: Participants]
  Never | 6
  Current | 12
  Former | 8
Alcohol use [Count of Participants; unit: Participants]
  Never | 4
  Current | 12
  Former | 10
Previous Tuberculosis (TB) diagnoses [Count of Participants; unit: Participants] — Population: participant may have had more than one occurrences of previous TB diagnosis and could select more than one category.
  Participants
    DS-TB | 7
    INH Mono-resistant TB | 2
    RIF mono-resistant TB | 15
    MDR-TB | 9
Screening smear microscopy for Acid Fast Bacilli (AFB) [Count of Participants; unit: Participants] — Detected acid-fast bacilli (AFB) by microscopic examination of clinical sputum specimens and cultures collected from participants. A quantitative grading system (WHO/IUATLD scaling system) was used to report the number of AFB observed in stained smears from concentrated sputum specimens, ranging from none seen to a 3+, depending on the amount of bacilli counted on microscopic examination.
  Participants
    No AFB seen | 6
    Scanty Positive | 4
    1+ | 3
    2+ | 3
    3+ | 10
Time to positivity at baseline [Mean (Standard Deviation); unit: Days] — The Time to Positivity (TTP) analysis is based on the number of participants who had a positive MGIT at baseline. One MGIT result had not been reported at the time the primary results were reported. N=21 in subsequent reports. Population: Only for those positive (MGIT) at baseline (between Day 1 and Week 4)
  Days
    number analyzed (Participants) | 21
    (all) | 9.9 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Change Form Baseline Total Sperm Count
Description: Change from baseline in total sperm number at 26 weeks of therapy. Total sperm count is calculated by multiplying the sperm cell concentration by the ejaculate volume.
Time Frame: Week 26
Population: Excludes participants not meeting definition of having received adequate treatment (80% of allocated doses) or with major protocol deviations including participants who did not satisfy entry criteria but were entered anyway; participants who developed withdrawal criteria during the study but were not withdrawn; and participants who received the wrong treatment or incorrect dose..
Measure: Mean (Standard Deviation); unit: 10^6 sperm cells/ejaculate
Arm/Group | BPaMZ
Number analyzed (Participants) | 22
10^6 sperm cells/ejaculate | 20 (97.3)

2. Secondary Outcome: Change From Baseline in Total Sperm Count at 12 Weeks
Description: Change from baseline in total sperm number at 12 weeks of therapy. Total sperm count is calculated by multiplying the sperm cell concentration by the ejaculate volume.
Time Frame: Baseline to Week 12
Population: Excludes participants not meeting definition of having received adequate treatment (80% of allocated doses)or with major protocol deviations including participants who did not satisfy entry criteria but were entered anyway; participants who developed withdrawal criteria during the study but were not withdrawn; and participants who received the wrong treatment or incorrect dose.
Measure: Mean (Standard Deviation); unit: 10^6 sperm cells/ejaculate
Arm/Group | BPaMZ
Number analyzed (Participants) | 22
10^6 sperm cells/ejaculate | 4.2 (56.8)

3. Secondary Outcome: Change From Baseline Total Sperm Count at 44 Weeks
Description: Change from baseline in total sperm number at 44 weeks (18 months post treatment completion). Total sperm count is calculated by multiplying the sperm cell concentration by the ejaculate volume.
Time Frame: Baseline through 44 weeks
Population: All enrolled participants who completed the 44-week visit.
Measure: Mean (Standard Deviation); unit: 10^6 sperm cells/ejaculate
Arm/Group | BPaMZ
Number analyzed (Participants) | 20
10^6 sperm cells/ejaculate | 4.4 (95.9)

4. Secondary Outcome: Luteinizing Hormone (LH)
Description: (LH) at baseline, 26, 44, and 78 weeks.
Time Frame: Baseline to Week 78
Population: Total assessable. (Excludes participants who were lost to follow-up or with missing data)
Measure: Median (Inter-Quartile Range); unit: IU/mL
Groups:
- BPaMZ Baseline; BPaMZ 26 Weeks; BPaMZ 44 Weeks; BPaMZ 78 Weeks: Participants will receive bedaquiline 200 mg once daily for 8 weeks then 100 mg once daily for 18 weeks together with pretomanid 200 mg + moxifloxacin 400 mg + pyrazinamide 1500 mg once daily (BPaMZ) for 26 weeks.
  Pretomanid: pretomanid 200 mg (once daily) for 26 weeks (with meal)
  Bedaquiline: bedaquiline 200 mg (once daily) for 8 weeks (with meal), then bedaquiline 100mg (once daily) for 18 weeks (with meal)
  moxifloxacin: moxifloxacin 400 mg (once daily) for 26 weeks (with meal)
  pyrazinamide: pyrazinamide 1500 mg (once daily) for 26 weeks (with meal)
Arm/Group | BPaMZ Baseline | BPaMZ 26 Weeks | BPaMZ 44 Weeks | BPaMZ 78 Weeks
Number analyzed (Participants) | 22 | 22 | 19 | 18
IU/mL | 5.8 [3.9 to 7.0] | 4.6 [3.5 to 5.6] | 3.6 [3.2 to 6.9] | 4.0 [3.5 to 6.2]

5. Secondary Outcome: FSH
Description: FSH at baseline, weeks 26, 44 and 78
Time Frame: Baseline to week 78
Population: Total assessable. (Excludes participants who were lost to follow-up or with missing data)
Measure: Median (Inter-Quartile Range); unit: IU/mL
Arm/Group | BPaMZ Baseline | BPaMZ 26 Weeks | BPaMZ 44 Weeks | BPaMZ 78 Weeks
Number analyzed (Participants) | 22 | 22 | 19 | 18
IU/mL | 6.6 [3.5 to 10.5] | 6.2 [3.7 to 9.7] | 5.2 [4.4 to 6.8] | 4.6 [2.6 to 5.8]

6. Secondary Outcome: Testosterone
Description: testosterone level at baseline, 26, 44 and 78 weeks.
Time Frame: Baseline to 78 weeks
Population: Total assessable. (Excludes participants who were lost to follow-up or with missing data)
Measure: Median (Inter-Quartile Range); unit: ng/dL
Arm/Group | BPaMZ Baseline | BPaMZ 26 Weeks | BPaMZ 44 Weeks | BPaMZ 78 Weeks
Number analyzed (Participants) | 22 | 22 | 19 | 18
ng/dL | 547 [444 to 688] | 600 [488 to 706] | 646 [499 to 820] | 615.5 [504 to 797]

7. Secondary Outcome: Inhibin B
Description: inhibin B at baseline, weeks 26, 44 and 78
Time Frame: Baseline to 78 weeks
Population: Total assessable. (Excludes participants who were lost to follow-up or with missing data)
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | BPaMZ Baseline | BPaMZ 26 Weeks | BPaMZ 44 Weeks | BPaMZ 78 Weeks
Number analyzed (Participants) | 21 | 21 | 20 | 18
pg/mL | 122 [72 to 155] | 137 [105 to 189] | 162.5 [96 to 194.5] | 172 [110 to 188]

ADVERSE EVENTS:
Time Frame: All adverse events (including Serious adverse events) listed in result's are treatment emergent; defined in this trial AEs which started or worsened on or after the first administration of BPaMZ up to and including last date scheduled study drug (up to 26 weeks) was administered plus 2 weeks following last treatment dose. .
Arm/Group | BPaMZ
All-Cause Mortality (participants affected / at risk) | 1/26
Serious Adverse Events (participants affected / at risk) | 2/26
Other Adverse Events (participants affected / at risk) | 21/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BPaMZ (N=26)
infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1)
hepatic enzyme increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BPaMZ (N=26)
constipation (Gastrointestinal disorders) | 3 (3)
diarrhoea (Gastrointestinal disorders) | 2 (2)
gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
haemorrhoids (Gastrointestinal disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 3 (3)
hypertransaminasaemia (Hepatobiliary disorders) | 2 (2)
conjunctivitis (Infections and infestations) | 2 (2)
lower respiratory infection (Infections and infestations) | 3 (3)
pneumonia (Infections and infestations) | 2 (2)
upper respiratory tract infection (Infections and infestations) | 4 (4)
aspartate aminotransferase increased (Investigations) | 2 (2)
blood potassium decreased (Investigations) | 3 (3)
blood uric acid increased (Investigations) | 2 (2)
gamma-glutamyltransferase increased (Investigations) | 2 (2)
hepatic enzyme increased (Investigations) | 2 (2)
decreased appetite (Metabolism and nutrition disorders) | 3 (3)
hyperuricaemia (Metabolism and nutrition disorders) | 4 (4)
hyponatraemia (Metabolism and nutrition disorders) | 3 (3)
arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
dizziness (Nervous system disorders) | 3 (3)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 5 (5)
dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
pruritus (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Principal Investigator shall not publish, present or use the Study Data for its own instruction, research or publication without the prior express written consent of Sponsor. Because the Study is funded, in whole or in part, by the Bill and Melinda Gates Foundation (the "Foundation"), all peer-reviewed published research relating to the Study must comply with the Foundation's Open Access Policy.

DOCUMENTS (2):
  • Study Protocol (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT04179500/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT04179500/SAP_001.pdf